CLINICAL TRIAL: NCT03982108
Title: Comparison of Repair Integrity and Functional Outcomes Between Knot-tying and Knotless Suture-bridge Arthroscopic Rotator Cuff Repair: a Prospective Randomized Clinical Trial
Brief Title: Comparison of Two Arthroscopic Rotator Cuff Repair Techniques: Knot-tying Versus Knotless Suture-bridge Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koray Sahin (Other)
Responsible Party: Sponsor-Investigator, Koray Sahin, Resident in orthopedics and traumatology department, Istanbul University
Organization: Istanbul University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IU-260133
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Rotator Cuff Tears; Rotator Cuff Injuries
Keywords: shoulder; rotator cuff tear; arthroscopic repair; suture-bridge technique; retear; knotless; knot-tying
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Knotless suture-bridge technique (Experimental): All participants in this arm will undergo an arthroscopic rotator cuff repair with knotless suture-bridge technique.
  Interventions: Procedure: Arthroscopic rotator cuff repair with knotless suture-bridge technique
- Knot-tying suture-bridge technique (Active Comparator): All participants in this arm will undergo an arthroscopic rotator cuff repair with knot-tying suture-bridge technique.
  Interventions: Procedure: Arthroscopic rotator cuff repair with knot-tying suture-bridge technique

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff repair with knotless suture-bridge technique — A posterior portal will be established to obtain adequate visualization and an anterior portal will be established through rotator interval as a working portal for diagnostic arthroscopy and debridement. Then additional portals will be established and preperation of tendon will be performed and a burr will be used for footprint preperation.
  After determination of proper anchor locations, required number of suture anchors will be inserted just lateral to articular margin depending on the tear size. Then limbs of sutures will be passed from the rotator cuff and will be used to create a suture bridge over the tendon. Then these limbs will be loaded to anchors which will form the lateral row without tying the suture limbs at the medial row. These lateral anchors will be inserted to adequate location, just lateral and distal to greater tuberosity with adequate suture-bridge tension over the rotator cuff.
  Arms: Knotless suture-bridge technique
Procedure: Arthroscopic rotator cuff repair with knot-tying suture-bridge technique — After the same preparation procedure as in knotless suture-bridge technique, required number of suture anchors will be inserted just lateral to articular margin depending on the tear size. Then limbs of sutures will be passed from the tendon and tied in a horizontal mattress suture pattern. After the establishment of medial row, suture limbs will be used to form a suture bridge over the tendon and will be loaded to lateral row anchors which then will be inserted lateral to greater tuberosity in a similar way to knotless repair technique.
  Arms: Knot-tying suture-bridge technique

SUMMARY:
Suture-bridge technique has been widely used for rotator cuff tears with many studies showing superior clinical results and lower failure rates compared to other techniques. This study aims to compare clinical outcomes and radiological integrity of arthroscopic rotator cuff repair between knot-tying and knotless suture-bridge techniques. The possibility of tendon strangulation and necrosis at the medial row when performing a suture-bridge technique may lead to retear and structural failure. In order to avoid this complication, the knots used at the medial row and their tension might be a factor to consider. Our hypothesis is that a knotless suture-bridge technique might avoid tendon strangulation thus might have lower retear rates.

DETAILED DESCRIPTION:
This study has been planned as a prospective randomized clinical trial. We used a completely computer-generated list in order to randomize all participants to receive one of two treatments (https://www.random.org/sequences/).

Rotator cuff tear diagnosis will be made by physical examination and magnetic resonance imaging. Participants who agree to be enrolled to study will be examined one day prior to surgery. Half of the participants will undergo an arthroscopic rotator cuff repair with knot-tying suture-bridge technique, while the other half will receive a knotless suture-bridge technique. All the surgeries will be performed by the same senior surgeon experienced in shoulder surgery under general anesthesia with participant in beach-chair position.

All participants will receive a standard postoperative rehabilitation program starting immediately after surgery with active elbow and passive shoulder exercises. The operated upper extremity will be placed in a sling for 6 weeks. Active-assisted exercises will be started at 6 weeks postoperatively.

Postoperative evaluations will be performed regularly at 2 weeks, 6 weeks, 3 months, 6 months, 12 months postoperatively and each following year. The results of last follow-up will be analyzed. To assess repair integrity and tendon healing, a postoperative magnetic resonance imaging scan will be performed to all participants at 6 months postoperatively. The results of prospective clinical follow-up data and radiological evaluation will be analyzed in order to compare clinical outcomes, failure rates and patterns of knot-tying and knotless suture-bridge arthroscopic rotator cuff repair techniques.

ELIGIBILITY:
Inclusion Criteria:

* Full thickness rotator cuff tear repaired by arthroscopic suture-bridge technique

Exclusion Criteria:

* Partial thickness rotator cuff tear
* Presence of a full thickness subscapularis tear that requires a repair
* History of a neurological disease
* Presence of severe glenohumeral or acromioclavicular arthritis
* Presence of a metal implant which prevents magnetic resonance imaging scan
* Tears repaired with other techniques
* Revision surgeries

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Sugaya classification of rotator cuff integrity | 6 months postoperatively
  This is a classification system described by Sugaya et al. which uses magnetic resonance imaging in order to evaluate tendon integrity after rotator cuff repair. Postoperative cuff integrity is classified into 5 categories: type I, sufficient thickness with homogenously low intensity; type II, sufficient thickness with partial high intensity; type III, insufficient thickness without discontinuity; type IV, presence of minor discontinuity; type V, presence of major discontinuity
Constant shoulder score | Change from baseline Constant shoulder score at 12 months
  This is a clinical functional assessment test used for shoulder disorders. The score consists of 4 sections: pain, activities of daily living, mobility and strength.

SECONDARY OUTCOMES:
Shoulder range of motion | Change from baseline range of motion at 12 months
  Shoulder abduction, forward flexion, external rotation, internal rotation and extension degrees measured by a goniometer
Visual analog scale for pain | Change from baseline visual analog scale for pain at 12 months
  A visual scale which classifies the intensity of pain between 0-10.
Retear patterns of rotator cuff tendons | 6 months postoperatively
  Retear patterns of rotator cuff tendons will be evaluated by using postoperative magnetic resonance images. Detected retears will be classified as type 1 (lateral) or type 2 (medial/musculotendinous) rotator cuff retears/failures.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ersen, M.D., Principal Investigator — Istanbul University Istanbul Medical Faculty
Locations (1):
- Istanbul University Istanbul Medical Faculty Department of Orthopedics and Traumatology, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angst F, Schwyzer HK, Aeschlimann A, Simmen BR, Goldhahn J. Measures of adult shoulder function: Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH) and its short version (QuickDASH), Shoulder Pain and Disability Index (SPADI), American Shoulder and Elbow Surgeons (ASES) Society standardized shoulder assessment form, Constant (Murley) Score (CS), Simple Shoulder Test (SST), Oxford Shoulder Score (OSS), Shoulder Disability Questionnaire (SDQ), and Western Ontario Shoulder Instability Index (WOSI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S174-88. doi: 10.1002/acr.20630. No abstract available. PMID 22588743
- [Background] Sugaya H, Maeda K, Matsuki K, Moriishi J. Functional and structural outcome after arthroscopic full-thickness rotator cuff repair: single-row versus dual-row fixation. Arthroscopy. 2005 Nov;21(11):1307-16. doi: 10.1016/j.arthro.2005.08.011. PMID 16325080
- [Result] Rhee YG, Cho NS, Parke CS. Arthroscopic rotator cuff repair using modified Mason-Allen medial row stitch: knotless versus knot-tying suture bridge technique. Am J Sports Med. 2012 Nov;40(11):2440-7. doi: 10.1177/0363546512459170. Epub 2012 Sep 21. PMID 23002202
- [Result] Kim KC, Shin HD, Cha SM, Park JY. Comparisons of retear patterns for 3 arthroscopic rotator cuff repair methods. Am J Sports Med. 2014 Mar;42(3):558-65. doi: 10.1177/0363546514521577. PMID 24585674
- [Result] Millett PJ, Espinoza C, Horan MP, Ho CP, Warth RJ, Dornan GJ, Katthagen JC. Predictors of outcomes after arthroscopic transosseous equivalent rotator cuff repair in 155 cases: a propensity score weighted analysis of knotted and knotless self-reinforcing repair techniques at a minimum of 2 years. Arch Orthop Trauma Surg. 2017 Oct;137(10):1399-1408. doi: 10.1007/s00402-017-2750-7. Epub 2017 Jul 26. PMID 28748291
- [Derived] Sahin K, Senturk F, Ersin M, Arzu U, Chodza M, Ersen A. Repair Integrity and Functional Outcomes Between Knot-Tying and Knotless Suture-Bridge Arthroscopic Rotator Cuff Repair: A Prospective Randomized Clinical Trial. Orthop J Sports Med. 2021 Apr 19;9(4):23259671211002482. doi: 10.1177/23259671211002482. eCollection 2021 Apr. PMID 33954223
- See also: Web site used for randomization of participants — https://www.random.org/sequences/